CLINICAL TRIAL: NCT02516085
Title: Improved Muscle Function in Duchenne Muscular Dystrophy Through L-Arginine and Metformin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Principal Investigator, Dirk Fischer, MD, University Hospital, Basel, Switzerland
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DMD01
Record Dates: First submitted 2015-08-03; First posted 2015-08-05 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-08

CONDITIONS: Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — Metformin; Arginine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- L-arginine and metformin (Experimental): 7.5 g L-arginine p.o. and 500 mg metformin p.o. per day (3x 2.5 g, respectively 3x 250 mg) for 16 weeks
  Interventions: Drug: Metformin; Drug: L-Arginine

INTERVENTIONS:
Drug: Metformin
Drug: L-Arginine

SUMMARY:
The purpose of the study is to show that the intake of L-arginine and metformin improves muscle function and delays disease progression in patients with Duchenne's muscular dystrophy.

DETAILED DESCRIPTION:
This is an investigator-initiated, open-label, single-center, proof-of-concept-study. The study medication consists of L-arginine and metformin. The duration of the study is 16 weeks and comprehends one screening and four study visits.

ELIGIBILITY:
Inclusion Criteria:

* Molecular diagnosis of DMD
* Patients 7 - 10 years of age at time of screening
* Ambulant

Exclusion Criteria:

* Previous (3 months or less) or concomitant participation in another therapeutic trial
* Use of L-arginine, L-citrulline or metformin within the last 3 months
* Known individual hypersensitivity to L-citrulline or metformin
* Other chronic disease or clinical relevant limitation of renal, liver, heart function according to discretion of the investigator

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2012-01; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Mean change of muscle metabolism | baseline to week 16
  mitochondrial protein expression analysis in muscular biopsies

SECONDARY OUTCOMES:
In vivo change of muscle metabolism | baseline to week 16
  indirect calorimetry, Dual-Energy X-Ray Absorptiometry, quantitative thigh muscle MRI, clinical score of muscle performance

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Fischer, MD, Principal Investigator — University of Basel, Children's Hospital

REFERENCES:
- [Derived] Hafner P, Bonati U, Erne B, Schmid M, Rubino D, Pohlman U, Peters T, Rutz E, Frank S, Neuhaus C, Deuster S, Gloor M, Bieri O, Fischmann A, Sinnreich M, Gueven N, Fischer D. Improved Muscle Function in Duchenne Muscular Dystrophy through L-Arginine and Metformin: An Investigator-Initiated, Open-Label, Single-Center, Proof-Of-Concept-Study. PLoS One. 2016 Jan 22;11(1):e0147634. doi: 10.1371/journal.pone.0147634. eCollection 2016. PMID 26799743